CLINICAL TRIAL: NCT06664177
Title: Comparison of the Postoperative Analgesic Efficacy of Quadratus Lumborum Block and Transversalis Fascia Block in Inguinal Hernia Surgery
Brief Title: Analgesic Efficacy of Quadratus Lumborum vs. Transversalis Fascia Block in Inguinal Hernia Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, SERPİL ŞEHİRLİOĞLU, principal invertigator, Gaziosmanpasa Research and Education Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: GaziosmanpasaTREH-FT-İH
Record Dates: First submitted 2024-10-27; First posted 2024-10-29 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Pain, Postoperative
Keywords: quadratus lumborum block; Transversalis Fascia Plane Block; inguinal hernia
MeSH Terms: conditions — Pain, Postoperative; Hernia, Inguinal

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anterior quadratus lumborum block (Active Comparator): The anterior QLB block will be applied on the operative side
  Interventions: Procedure: Anterior Quadratus Lumborum Block (QLB)
- transversalis fascia group (Active Comparator): the Transversalis Fascia Block will be applied on the operative side
  Interventions: Procedure: Transversalis Fascia Plane Block

INTERVENTIONS:
Procedure: Transversalis Fascia Plane Block — In the Transversalis Fascia Block group, the same procedure will be followed as in the Quadratus Lumborum block group, with the ultrasound probe being placed in the same location, and the same in-plane technique will be applied with a 22G 100 mm peripheral block needle. After hydrodissection, 20 mL of 0.25% bupivacaine will be injected slowly in the same manner.
  Arms: transversalis fascia group
Procedure: Anterior Quadratus Lumborum Block (QLB) — In the Quadratus Lumborum block group, in the lateral decubitus position, a convex ultrasound probe will be sterilely placed in the subcostal area and above the iliac crest. The quadratus lumborum and psoas major muscles, as well as the L4 vertebra's transverse process, will be visualized. Using the in-plane technique and a 22G 100 mm peripheral block needle, the placement will first be identified through hydrodissection in the subfascial area between the quadratus lumborum and psoas major muscles. After localization, 20 mL of 0.25% bupivacaine will be injected slowly, aspirating every 5 cc, while visualizing the local anesthetic pushing the fascia in the ultrasound image.
  Arms: anterior quadratus lumborum block

SUMMARY:
It is planned to compare the postoperative analgesic efficacy of the Transversalis Fascia Plane Block and the anterior Quadratus Lumborum Block in elective inguinal hernia surgeries.

DETAILED DESCRIPTION:
It is planned to compare the postoperative analgesic efficacy of the Transversalis Fascia Plane Block and the anterior Quadratus Lumborum Block in elective open inguinal hernia surgeries.

Primary Objective: Our primary aim is to compare and evaluate the time to first rescue analgesic requirement after the application of anterior Quadratus Lumborum Block and Transversalis Fascia Plane Block in patients undergoing elective open inguinal hernia surgeries under spinal anesthesia.

Secondary Objectives:

To compare the total analgesic consumption in the first 24 hours postoperatively.

To compare the Numeric Rating Scale (NRS) values (at rest and dynamic) of patients at postoperative follow-ups at 2, 4, 8, 12, and 24 hours.

To compare postoperative side effects such as nausea and vomiting. In trunk blocks, local anesthetic is applied to the interfascial area between the anterior abdominal wall or back muscles. Due to the lack of blood circulation and vascularization in the interfascial area, the absorption of local anesthetics is slow, allowing for prolonged analgesic effects. For this reason, trunk blocks are used as part of multimodal analgesia. The effectiveness of trunk blocks can vary based on the patient's structural anatomical differences and previous surgeries, but an average analgesic effect of 8-12 hours is typically observed. Sometimes, analgesic effects have been reported to last up to 24 hours.

Pain that arises from elective laparoscopic inguinal hernia surgeries can negatively impact postoperative immobilization, atelectasis, pneumonia due to atelectasis, and prolonged hospital stays. Due to the side effects associated with opioid medications used for postoperative analgesia, such as nausea, vomiting, itching, constipation, and dependency, non-opioid analgesic medications and regional techniques are used as part of multimodal analgesia to reduce opioid use.

Quadratus Lumborum and Transversalis Fascia Blocks can be safely and easily performed, especially in lower abdominal surgery, due to advancements in trunk blocks and ultrasound technology in recent years.

This study aims to evaluate the postoperative analgesic efficacy of Quadratus Lumborum Blocks and Transversalis Fascia Blocks administered to patients undergoing elective inguinal hernia surgery. The Transversalis Fascia Block can be utilized in lower abdominal surgeries by blocking the ilioinguinal, iliohypogastric nerves, and the T12 intercostal nerve. The Quadratus Lumborum Block provides analgesic efficacy in the T7-L2 dermatomal area.In patients planned for elective laparoscopic inguinal hernia surgery, informed consent was obtained after detailed information was provided. The patients were randomly divided into two groups using closed envelope randomization: the anterior Quadratus Lumborum Block group and the Transversalis Fascia Block group.

All patients will be taken to the block room after the surgery. All blocks will be performed under ultrasound guidance by the same anesthesia specialist while the patients are in the lateral decubitus position, with the surgical sites facing up.

In the Quadratus Lumborum block group, in the lateral decubitus position, a convex ultrasound probe will be sterilely placed in the subcostal area and above the iliac crest. The quadratus lumborum and psoas major muscles, as well as the L4 vertebra's transverse process, will be visualized. Using the in-plane technique and a 22G 100 mm peripheral block needle, the placement will first be identified through hydrodissection in the subfascial area between the quadratus lumborum and psoas major muscles. After localization, 20 mL of 0.5% bupivacaine will be injected slowly, aspirating every 5 cc, while visualizing the local anesthetic pushing the fascia in the ultrasound image.

In the Transversalis Fascia Block group, the same procedure will be followed as in the Quadratus Lumborum block group, with the ultrasound probe being placed in the same location, and the same in-plane technique will be applied with a 22G 100 mm peripheral block needle. After hydrodissection, 20 mL of 0.5% bupivacaine will be injected slowly in the same manner.

All patients will be monitored for 30 minutes in the block room after the block application.

All patients will receive anesthesia using the same technique under spinal anesthesia with bupivacain 12 mg intratechal space before surgery. At the end of the operation, all patients will receive intravenous 1g of paracetamol for postoperative analgesia. Routine extubation will be performed, and patients will be sent to the ward after recovery.

Postoperative analgesia for patients was planned as paracetamol 4x1g. Patients will be followed up by a different blinded anesthesia assistant from the one who performed the block at 2, 4, 8, 12, and 24 hours. The first rescue analgesia times, NRS scores (evaluated on a scale of 1 to 10, where 0 means no pain and 10 means very severe pain), postoperative side effects, and total analgesic amounts used in 24 hours will be recorded.

In postoperative follow-ups, for patients with NRS scores greater than 3, intravenous ibuprofen will be planned as rescue analgesia in the ward. If pain does not resolve within 30 minutes, dexketoprophen 50 mg IV will be planned.

In trunk blocks, blocking the thoracoabdominal nerves that travel between the fascia with local anesthetics is thought to provide analgesia during the postoperative period, increasing patient comfort, reducing postoperative opioid consumption and dependency, facilitating early mobilization, shortening the hospital stay, and minimizing opioid side effects.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65
* ASA Classification 1-2

Exclusion Criteria:

* Allergy to local anesthetics
* Presence of infection at the procedure site
* BMI > 35 kg/m²
* Bleeding disorders or anticoagulant use
* Chronic analgesic or opioid use
* Mental or psychiatric disorders
* ASA Classification 3-4 patients(Severe COPD, history of cerebrovascular events, liver and kidney disease will be excluded from the study.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
time to first rescue analgesic requirement. | 24 hour
  Our primary aim is to compare and evaluate the time to first rescue analgesic requirement after the application of anterior Quadratus Lumborum Block and Transversalis Fascia Plane Block in patients undergoing elective inguinal hernia surgeries under spinal anesthesia.

SECONDARY OUTCOMES:
Total Opioid Consumption | 24 hour
  To compare the total analgesic consumption in the first 24 hours postoperatively.
To compare the NRS (Numering rating scale) values (resting and dynamic) at 2. 4. 8. 12 . 24. hours in the postoperative follow-up of the patients | 24 hour
  Assessed at various time points to quantify pain intensity at rest and during movement. The Numerical Rating Scale (NRS) is a pain assessment tool where patients rate their pain from 0 (no pain) to 10 (worst pain).

CONTACTS AND LOCATIONS:
Overall Officials: Serpil Sehirlioglu, MD, Principal Investigator — Gaziosmanpasa Research and Education Hospital
Locations (1):
- Gaziosmanpasa Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data associated with the paper are not publicly available but are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: always
Access Criteria: drserpilsahin@gmail.com

REFERENCES:
- [Result] Abdelbaser I, Mageed NA, El-Emam EM, ALseoudy MM, Elmorsy MM. Preemptive analgesic efficacy of ultrasound-guided transversalis fascia plane block in children undergoing inguinal herniorrhaphy: a randomized, double-blind, controlled study. Korean J Anesthesiol. 2021 Aug;74(4):325-332. doi: 10.4097/kja.20601. Epub 2020 Dec 14. PMID 33307633
- [Result] Samerchua A, Leurcharusmee P, Panichpichate K, Bunchungmongkol N, Wanvoharn M, Tepmalai K, Khorana J, Chantakhow S. A Prospective, randomized comparative study between ultrasound-guided posterior quadratus lumborum block and ultrasound-guided ilioinguinal/iliohypogastric nerve block for pediatric inguinal herniotomy. Paediatr Anaesth. 2020 Apr;30(4):498-505. doi: 10.1111/pan.13837. Epub 2020 Feb 21. PMID 32030845
- [Result] Ahmed A, Fawzy M, Nasr MAR, Hussam AM, Fouad E, Aboeldahb H, Saad D, Osman S, Fahmy RS, Farid M, Waheb MM. Ultrasound-guided quadratus lumborum block for postoperative pain control in patients undergoing unilateral inguinal hernia repair, a comparative study between two approaches. BMC Anesthesiol. 2019 Oct 17;19(1):184. doi: 10.1186/s12871-019-0862-z. PMID 31623572